CLINICAL TRIAL: NCT03570606
Title: A Multi-centred, Post-market Clinical Follow-up Study of Synthetic Bone Graft Substitutes for Use in Orthopaedic and Spinal Applications.
Brief Title: Clinical Study of Bone Graft Substitutes in Orthopaedic and Spinal Applications.
Acronym: ROSA
Status: Active, not recruiting | Type: Observational
Sponsor: Ceramisys Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ROSA01
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Bone Deformity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (7):
- HA Paste in Spine: Evaluation of HA Paste in spinal fusion procedures
  o Spinal cage filling
  Interventions: Device: bone graft substitute
- HA Paste in long bone & extremities: Evaluation of HA Paste in long bone and extremity group:
  * Filling bone defects after cyst removal
  * Filling distal radius fractures
  * Filling defects such as tibial plateau fractures
  * Filling defects created by osteotomy procedures
  Interventions: Device: bone graft substitute
- Granulated Paste in Spine: Evaluation of Granulated Paste in spinal fusion procedures
  o Spinal cage filling
  Interventions: Device: bone graft substitute
- Granulated Paste in long bone & extremities: Evaluation of Granulated Paste in long bone and extremity group:
  * Filling bone defects after cyst removal
  * Filling distal radius fractures
  * Filling defects such as tibial plateau fractures
  * Filling defects created by osteotomy procedures
  Interventions: Device: bone graft substitute
- Granules in Spine: Evaluation of Granules in spinal fusion procedures
  o Spinal cage filling
  Interventions: Device: bone graft substitute
- Granules in long bone & extremities: Evaluation of Granules in long bone and extremity group:
  * Filling bone defects after cyst removal
  * Filling distal radius fractures
  * Filling defects such as tibial plateau fractures
  * Filling defects created by osteotomy procedures
  Interventions: Device: bone graft substitute
- Block in long bone & extremities: Evaluation of Blocks in long bone and extremity group:
  o High tibial osteotomies with fixation
  Interventions: Device: bone graft substitute

INTERVENTIONS:
Device: bone graft substitute — orthopaedic or spine bony defects

SUMMARY:
This is an observational, prospective, non-randomised, multi-centred post market clinical follow-up study to compile real world clinical data on safety and efficacy of the synthetic bone graft substitutes in a commercial clinical setting in long bone and extremity defects and in spinal fusion procedures.

ELIGIBILITY:
Inclusion Criteria:

Long Bone and Extremity Indications: patients requiring bone grafting after post-traumatic or surgically created bone defects afflicting the long bones and extremities.

Spine Indication: patients with degenerative disc disease or trauma who require spinal fusion of 1 or more vertebral bodies and where conservative treatment has been unsuccessful.

Patients who are willing and capable of providing informed consent, participating in all testing associated with this clinical investigation at an approved clinical investigational center;

Exclusion Criteria:

Patients who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the patient is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance should be brought to the attention of the sponsor to determine eligibility.

Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon physician's discretion); The subject is unable or not willing to complete follow-up visits and examination for the duration of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male or female 18-80 meeting the inclusion criteria, provided no exclusion criteria are met:
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary endpoints will be successful radiographic bone repair. | 12 months
  Bone formation and material resorption, observable by x-ray/MRI

CONTACTS AND LOCATIONS:
Locations (7):
- United Kingdom (7):
  - Doncaster & Bassetlaw Teaching Hospitals NHS Foundation Trust, Doncaster, South Yorkshire
  - Sandwell and West Birmingham NHS Trust of City Hospital, Birmingham
  - The Royal Orthopaedic Hospital NHS Foundation Trust, Birmingham
  - Northumbria Healthcare NHS Foundation Trust, North Shields
  - Salford Royal NHS Foundation Trust, Salford
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent
  - Taunton and Somerset NHS Foundation Trust, Taunton

IPD SHARING:
Plan to Share IPD: No